CLINICAL TRIAL: NCT02248896
Title: Antihypertensive Medications and the Risk of Sepsis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.590
Record Dates: First submitted 2014-09-24; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hypertensive patients: Hypertensive patients or patients treated with antihypertensive drugs with linked GPRD and hospital episodes statistics database (HES) data
  Interventions: Drug: Telmisartan; Drug: Other angiotensin-receptor blockers (ARBs); Drug: Angiotensin-converting enzyme inhibitors (ACEIs); Drug: Other major antihypertensive medication classes

INTERVENTIONS:
Drug: Telmisartan
Drug: Other angiotensin-receptor blockers (ARBs)
Drug: Angiotensin-converting enzyme inhibitors (ACEIs)
Drug: Other major antihypertensive medication classes — e.g. beta-blockers, calcium channel blockers (CCBs), diuretics

SUMMARY:
The primary objective of this study was to assess whether there is an increased risk of sepsis with the use of telmisartan compared with other ARBs and with the other major antihypertensive classes, including ACEIs, beta-blockers, CCBs and thiazide diuretics. A secondary objective was to assess whether the use of ARBs and ACEIs, compared with the other three major antihypertensive classes and with untreated hypertension, is associated with an increased risk of sepsis. A third objective was to evaluate whether the use of telmisartan compared with other ARBs, ACEIs and other major antihypertensive classes is associated with an increased risk of worse outcomes due to sepsis, in particular acute kidney injury and death

ELIGIBILITY:
Inclusion Criteria:

- Patients, 18 years or older, with at least two-year follow-up in United Kingdom's general practice research database (GPRD), who had a diagnosis of or treatment for hypertension

Exclusion Criteria:

- Sepsis, chronic renal failure or on dialysis in the two-year period prior to cohort entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of, or treatment for hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1129062 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Occurence of sepsis, including severe sepsis | Up to 9 years and 5 months
  Severe sepsis defined as cases that develop renal failure or die within 30 days